CLINICAL TRIAL: NCT05656118
Title: Safety and Efficacy of Paclitax Drug Coated Balloon Catheter (Genoss® DCB) in Patients With Coronary In-stent Restenosis (ISR): A Prospective, Multi-center, Observational Study (GENISPIRE Registry)
Brief Title: Safety and Efficacy of Paclitax Coated Balloon in Patients With Coronary In-stent Restenosis (ISR)
Acronym: GENISPIRE
Status: Active, not recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Deok-Kyu Cho, Professor, Department of Cardiology, Yongin Severance Hospital, Yonsei University College of Medicine, Yonsei University
Other Study IDs: 9-2022-0063
Record Dates: First submitted 2022-12-11; First posted 2022-12-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: In-stent Restenosis
Keywords: In-stent Restenosis; Drug-coated balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paclitaxel Coated Balloon: Patients treated with Genoss® DCB in patients with coronary artery in-stent restenosis (ISR)
  Interventions: Device: Genoss® DCB

INTERVENTIONS:
Device: Genoss® DCB — Paclitaxel coated balloon with a shellac plus vitamin E excipient

SUMMARY:
The purpose of this observational study was to evaluate the long-term efficacy and safety of a paclitaxel-coated balloon catheter in coronary in-stent restenosis (ISR) patients.

The primary endpoint was target lesion failure (TLF, a composite of cardiac death, target-vessel MI, or target lesion revascularization) at 12 months.

DETAILED DESCRIPTION:
260 subjects treated with a paclitaxel-coated balloon (Genoss® DCB) in patients with coronary in-stent restenosis (ISR) will be recruited and followed up to 12 months.

All enrolled patients treated with Genoss DCB in patients with coronary in-stent restenosis (ISR) will be included in the analysis unless there is a valid reason or rationale for it, and the final statistical analysis will follow the intention-to-treat (ITT) principle as assigned. Standard descriptive statistics will be used for patient baseline characteristics, lesions, procedures, and clinical event outcomes. Categorical variables will be presented as percentages and numbers and compared using chi-square or Fisher's exact test. Continuous variables will appear as mean, standard deviation or median, and interquartile range, and will be compared with Student's T-test or Wilcoxon rank sum test, and the normal value of the standard variable distribution will be predicted through histogram, skewness, kurtosis, and Kolmogorov Smirnov one sample test.

ELIGIBILITY:
Inclusion Criteria:

① Age ≥18 years old.

② Patients treated with Genoss® DCB in coronary artery In-stent restenosis (ISR) patients.

③ Patients who can understand the purpose of the study and voluntarily participate in and sign informed consent.

Exclusion Criteria:

* A woman who is pregnant, lactating, or planning a pregnancy. ② Patients who are scheduled for surgery requiring discontinuation of antiplatelet drugs within 12 months.

  * Patients with life expectancy less than 1 year.

    * Patients with cardiogenic shock and are predicted to have a low survival rate based on medical judgment.

      * Patients participating in a medical device randomized controlled trials. ⑥ Patients who, in the judgment of the investigator, are not suitable for this clinical study or may increase the risks associated with participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects treated with a paclitaxel-coated balloon (Genoss® DCB) in patients with coronary in-stent restenosis (ISR)
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Targeted lesion failure | 12 months
  A composite of cardiac death, target-vessel MI, or target lesion revascularization

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  A composite of all-cause death, MI, or revascularization
All-cause death | 12 months
  All-cause death and cardiac death
Any MI | 12 months
  Any MI and target vessel MI
Any revascularization | 12 months
  Any revascularization and ischemic driven target lesion revascularization
Major bleeding events, BARC 3, 5 | 12 months
  A composite rate of major bleeding events, BARC 3, 5
Any Stroke | 12 months
  Ischemic or hemorrhagic stroke
Any stent thrombosis | 12 months
  Definite or probable stent thrombosis (acute, subacute, late)

CONTACTS AND LOCATIONS:
Overall Officials: Deok-Kyu Cho, MD, Principal Investigator — Yongin Severance Hospital, Yonsei University
Locations (10):
- South Korea (10):
  - Kosin University Gospel Hospital, Busan, Busan
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - National Health Insurance Service Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Yongin Severance Hospital, Yonsei University, Yongin-si, Gyeonggi-do
  - Kyungpook National University College Hospital, Daegu, Gyeongsangnam-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Korea University ANAM Hospital, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No
The data set is available from the the corresponding author upon reasonable request.